CLINICAL TRIAL: NCT01105481
Title: Amisulpride Augmentation Therapy for Clozapine-resistant Schizophrenic Patients: A 14-week Randomized, Double-blind and Placebo-controlled Trial
Brief Title: Amisulpride Augmentation Therapy for Clozapine-resistant Schizophrenic Patients
Acronym: M1106
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Dr. Sheng-Chang Wang, Division of Mental Health and Addiction Medicine, National Health Research Instiutes, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M1106
Record Dates: First submitted 2010-03-31; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Treatment-resistant Schizophrenia
Keywords: treatment-resistant schizophrenia; clozapine; amisulpride
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amisulpride add-on (Experimental)
  Interventions: Drug: Amisulpride add-on
- placebo add-on (Placebo Comparator)
  Interventions: Drug: Placebo add-on

INTERVENTIONS:
Drug: Amisulpride add-on — At the beginning of the treatment phase (day 1), subjects in the combination treatment group will be started with adjunctive amisulpride, with a starting dose of 200 mg per day. Amisulpride is planned to increase to 400 mg/day on day 8, 600mg/day on day 15 and 800 mg/day on day 22, according to the subjects' responses and tolerability. All of the add-on amisulpride will be provided to subjects at night. To permit dose adjustment and ensure double-blind procedure, 200mg amisulpride is packed in capsules identical to those used for the placebo.
  Arms: amisulpride add-on
Drug: Placebo add-on — For subjects randomly allocated to the placebo treatment group, they will be added with one capsule of placebo from Day 1. On Day 8, Day 15 and Day 22, the placebo will be increased to 2, 3 and 4 capsules, respectively. and adjunctive amisulpride, with a starting dose of 200 mg per day. Amisulpride is planned to increase to 400 mg/day on day 8, 600mg/day on day 15 and 800 mg/day on day 22, according to the subjects' responses and tolerability. To permit dose adjustment and ensure double-blind procedure, 200mg amisulpride is packed in capsules identical to those used for the placebo.
  Arms: placebo add-on

SUMMARY:
This study includes two main components: the first screening phase and the second clinical intervention phase. During the screening phase, subjects with poor response to clozapine are carefully evaluated by chart-review and clinical assessment. Via chart-review, clinical data of diagnosis, disease course and previous treatment outcome, and concomitant psychotropic agents are obtained. Clinical phenomenology, including psychopathology, psychotic and mood symptoms severity and side effect of psychotropic medication are assessed by clinical interview and observation, which are conducted by experienced clinicians. Blood sample will be also obtained from the subjects for measuring the baseline clozapine drug level and extracting DNA for further analysis. Subjects fulfilling the criteria of treatment-resistant schizophrenia with poor response to adequate dose and duration of clozapine treatment are eligible for the clinical trial phase of 14-week randomized, placebo-controlled amisulpride add-on study. In this phase, subjects are randomly allocated to amisulpride augmentation treatment group and placebo treatment group. Subjects in the former group will receive clozapine and amisulpride combination treatment, while in the latter group will receive clozapine and placebo. Outcomes of clinical efficacy and safety are carefully evaluated by experienced and well-trained research stuffs in the 14 weeks of clinical study period.

All of the above studies will be conducted in four hospitals, including DOH Bali Psychiatric Hospital, DOH Tao-yan Psychiatric hospital, and the Ju-Shang Psychiatric Hospital. Subjects will be recruited from the chronic in-patient settings from these three hospitals.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosed schizophrenic patients;
* Age between 18 and 60;
* Before treatment with clozapine, documented treatment failure of two antipsychotics for an adequate duration of 6 weeks and in a sufficient dose of 600 mg/day of chlorpromazine equivalents;
* Documented failure to show a satisfactory clinical response to an adequate clozapine treatment, defined as at least clozapine 300 mg/day for 3 months or a plasma drug level of 350ng/ml;
* At least moderately ill, defined as with a Clinical Global Impression (CGI) greater than 4 or PANSS total score greater than 75;
* Persistent positive psychotic symptoms, with rating scores of moderate or worse on at least two of four positive symptom items (delusion, conceptual disorganization, hallucinatory behavior, and suspiciousness/persecution) on Positive and Negative Syndrome Scale (PANSS);

Exclusion Criteria:

* Patients with concomitant treatment with lithium, anti-convulsants, antidepressants and other antipsychotic medication ;
* Patients with underlying severe medical illness, such as cardiovascular disease, cerebrovascular disease, bone marrow suppression or epilepsy;
* Patients with comorbid diagnosis of substance dependence;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale(PANSS) total score change | 12 wks after treatment
  The change from baseline of the Positive and Negative Symptom Scale (PANSS) total score.

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) positive-symptom subscale score | 12 wks after treatment
  The change from baseline of the Positive and Negative Symptom Scale (PANSS) positive-symptom subscale score (sum of item P1 to P7)
Positive and Negative Symptom Scale (PANSS) negative-symptom subscale score | 12 wks after treatment
  The change from baseline of the Positive and Negative Symptom Scale (PANSS) negative-symptom subscale score (sum of item N1 to N7)
Positive and Negative Symptom Scale (PANSS) general psychopathology score | 12 wks after treatment
  The change from baseline of the Positive and Negative Symptom Scale (PANSS) general psychopathology subscale score (sum of item G1 to G14)
Clinical Global Impressions (CGI) scale score | 12 wks after treatment
  The change from baseline of the Clinical Global Impressions (CGI) scale score
Brief Psychotic Rating Scale (BPRS) total score | 12 wks after treatment
  The change from baseline of the Brief Psychotic Rating Scale (BPRS) score

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chang Wang, M.D.,M.Sc., Principal Investigator — National Health Research Institutes, Taiwan
Locations (2):
- Taiwan (2):
  - Bali Psychiatric Center, Taipei County
  - Departments of Psychiatry, Tao-yuan Psychiatric Center, Taoyuan District